CLINICAL TRIAL: NCT00804726
Title: A Prospective, Open-label, Monocular Feasibility Clinical Evaluation of the Bausch & Lomb Akreos MI Five-O Accommodating Intraocular Lens.
Brief Title: Evaluation of the Safety and Effectiveness of the Akreos MI Five-0 Intraocular Lens.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Test lens did not meet near visual efficacy endpoints
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 580
Record Dates: First submitted 2008-12-08; First posted 2008-12-09 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2014-01

CONDITIONS: Cataract
Keywords: Cataract extraction; Phacoemulsification
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Akreos MI Five-O (Experimental): Accommodating intraocular lens
  Interventions: Device: Akreos MI Five-O

INTERVENTIONS:
Device: Akreos MI Five-O — Small incision cataract surgery with phacoemulsification cataract extraction and Akreos MI Five-O IOL surgical implantation

SUMMARY:
The objective of this 12-month clinical investigation is to evaluate the safety and effectiveness of the Bausch & Lomb Akreos MI Five-O intraocular lens (IOL). Effectiveness will be shown through the demonstration of accurate distance correction and safety will be demonstrated through the monitoring of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a clinically documented diagnosis of age-related cataract.
* Subjects must have clear intraocular media other than cataract.
* Subjects must be undergoing primary in-the-bag intraocular lens implantation for the correction of aphakia following continuous curvilinear anterior capsulotomy and phacoemulsification cataract extraction.

Exclusion Criteria:

* Subjects with any anterior segment pathology for which extracapsular phacoemulsification cataract surgery would be contraindicated.
* Subjects with diagnosis of degenerative visual disorder.
* Subjects who have any inflammation or edema (swelling) of the cornea.
* Subjects with immunodeficiency disorders.
* Subjects who have had previous intraocular surgery in the study eye.
* Subjects with incomplete/damaged zonule, or with conditions associated with increased risk of zonular rupture.
* Subjects with chronic use of systemic steroids or immunosuppressive medications.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-11; Primary Completion 2010-05 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Visual acuity | 5 visits up to 420 days
  Uncorrected distance visual acuity Best corrected distance visual acuity Uncorrected near visual acuity Uncorrected intermediate visual acuity Near visual acuity with distance best correction

SECONDARY OUTCOMES:
Visual acuity | 5 visits up to 420 days
  Best corrected near Visual acuity Intermediate visual acuity with distance best correction Subjective near point of accommodation (push down test)

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Allmeier, PhD, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Augenzentrum Maus Wolfsstr 16, Cologne, Germany